CLINICAL TRIAL: NCT05075616
Title: A Retrospective Analysis of Percutaneous Endoscopic Gastrostomy Application Experiences to Geriatric Patients in Palliative Care Unit
Brief Title: A Retrospective Analysis of Percutaneous Endoscopic Gastrostomy Experiences
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Murat Ferhat Ferhatoglu, Assistant Professor, Okan University
Other Study IDs: 08.09.2021/141
Record Dates: First submitted 2021-10-02; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Nutrition Disorders; Gastrostomy
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Percutaneous endoscopic gastrostomy — Percutaneous endoscopic gastrostomy (PEG) is a minimally-invasive endoscopic procedure that creates a passage from the patient's stomach to the abdominal wall via a feeding tube and provides a means of feeding if oral intake is not adequate.

SUMMARY:
The application of PEG in geriatric-palliative care has not been well discussed. With the development of endoscopic procedures and PEG devices, we can perform this minimally invasive method more safely, even in challenging cases. We should discuss the indications of PEG in the field of palliative care of geriatric patients.

The presented study evaluated geriatric (> 65-year-old) palliative care patients to whom PEG applied at our institution.

DETAILED DESCRIPTION:
Palliative care is a treatment method that focuses on the patient and patient's family, aims to minimize the complaints caused by chronic diseases that cannot be treated, and increases life quality. The National Institute for Health and Care Excellence defines palliative care as; the active, holistic care of patients with an advanced progressive illness. Management of pain and other symptoms and providing psychological, social, and spiritual support is paramount. Anorexia, weight loss, and sarcopenia are highly visible and distressing reminders of the life-limiting disease's influence on patients who require palliative care. Given this multifaceted and significant role, it is not unexpected that nutritional treatment method choices can be challenging.

Percutaneous endoscopic gastrostomy (PEG) is a minimally-invasive endoscopic procedure that creates a passage from the patient's stomach to the abdominal wall via a feeding tube and provides a means of feeding if oral intake is not adequate. This safe and effective minimally-invasive option has been utilized in medical practice for over 40 years. PEG has advantages such as being minimally invasive, causing a low rate of complications and morbidity, and providing a long-lasting and safe feeding route. It is currently the chosen procedure for medium- and long-term enteral feeding in cases who need palliative care.

The application of PEG in geriatric-palliative care has not been well discussed. With the development of endoscopic procedures and PEG devices, we can perform this minimally invasive method more safely, even in challenging cases. We should discuss the indications of PEG in the field of palliative care of geriatric patients.

The presented study evaluated geriatric (> 65-year-old) palliative care patients to whom PEG applied at our institution.

ELIGIBILITY:
Inclusion Criteria:

- We retrospectively assessed the medical datum of PEG applied >65-year-old patients at our institution between December 2017 and March 2021 in our clinic.

Exclusion Criteria:

* We excluded the patients who were not treated in our palliative care center.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively assessed the medical data of PEG applied >65-year-old patients at our institution between December 2017 and March 2021. And, we excluded the patients who were not treated in our palliative care center. Table 1. shows the contraindications for PEG placement.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Weight and body mass index changes | 30 days
  Evaluation of weight and body mass index changes after Percutaneous endoscopic gastrostomy tube application

CONTACTS AND LOCATIONS:
Overall Officials: Murat Ferhat Ferhatoglu, MD, Study Director — Okan
Locations (2):
- Turkey (Türkiye) (2):
  - Okan University Hospital, Istanbul
  - Okan University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
Th excel file including study data will be shared.